CLINICAL TRIAL: NCT07342322
Title: A Prospective, Multicenter, Open-label, Single-arm Phase II Clinical Study Evaluating the Efficacy and Safety of Spatially Fractionated Radiotherapy Combined With the PraG Strategy for the Treatment of Soft Tissue Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-K0608
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Sarcoma (STS)
MeSH Terms: conditions — Sarcoma | interventions — toripalimab; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SFRT + PraG (Experimental)
  Interventions: Drug: Spatially Fractionated Radiation Therapy Combined with Toripalimab and Human Granulocyte-Macrophage Colony-Stimulating Factor for Injection

INTERVENTIONS:
Drug: Spatially Fractionated Radiation Therapy Combined with Toripalimab and Human Granulocyte-Macrophage Colony-Stimulating Factor for Injection — 1. Spatially Fractionated Radiation Therapy:
     1. High-dose area: 500-800 cGy × 3 fractions
     2. Fraction interval: 1 session of radiotherapy per day, with 3 sessions per cycle
     3. High-dose area coverage: 40-60% of the irradiated field area
  2. Toripalimab:
     1. Dose: 3 mg/kg
     2. Frequency: Every 2-3 weeks
     3. Administration timing: Within one week after the completion of radiotherapy
  3. Human Granulocyte-Macrophage Colony-Stimulating Factor for Injection:
     1. Dose: 100-200 µg
     2. Frequency: Once daily
     <!-- -->
     1. Administration timing: Starting on the day of radiotherapy, to be used continuously for one week

SUMMARY:
The primary objective of this clinical trial is to evaluate the efficacy and safety of spatially fractionated radiotherapy combined with the PraG strategy in the treatment of soft tissue sarcoma (STS). The main questions it aims to answer are:

1. Can spatially fractionated radiotherapy combined with the PraG strategy improve the clinical prognosis of patients?
2. What medical adverse events and clinical problems will participants encounter during the treatment with spatially fractionated radiotherapy combined with the PraG strategy? Researchers will administer a combined therapeutic regimen consisting of spatially fractionated radiotherapy, Toripalimab, recombinant human granulocyte-macrophage colony-stimulating factor injection, and Thymalfasin injection to enrolled patients, so as to observe the efficacy and safety of this therapeutic strategy for soft tissue sarcoma.

Participants will:

1. The treatment will be divided into two major phases: the radiotherapy phase and the immunotherapy phase, with concomitant immunomodulatory supportive therapy administered throughout the entire treatment course.
2. The total duration of treatment will last for 1 year starting from the first dose of medication, with regular clinical evaluations conducted according to the individual disease characteristics of each patient.
3. Participants will receive daily oral administration of ABC or placebo for a consecutive 4 months.
4. Routine follow-up examinations will be performed at an interval of 8/12 weeks.
5. Clinical symptoms, imaging indicators, biochemical parameters and survival status of all participants will be systematically recorded and documented throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, both genders are eligible.
2. Pathological Diagnosis: Histologically confirmed soft tissue sarcoma, including but not limited to:

   * Undifferentiated pleomorphic sarcoma
   * Liposarcoma
   * Leiomyosarcoma
   * Synovial sarcoma
   * Fibrosarcoma
   * Other high-grade soft tissue sarcomas
3. Disease Stage:

   * Locally advanced, unresectable soft tissue sarcoma, or
   * Recurrent or metastatic soft tissue sarcoma
4. Prior Therapy:

   * Prior surgery, radiotherapy, or chemotherapy is allowed.
   * At least 4 weeks since the last anti-tumor treatment.
   * Prior treatment-related toxicities have resolved to ≤Grade 1 (except alopecia).
5. Measurable Disease: At least one measurable lesion according to RECIST 1.1 criteria.
6. Performance Status: ECOG performance status score of 0-2.
7. Life Expectancy: ≥3 months.
8. Organ Function:

   * Hematology: Hemoglobin ≥50 g/L, absolute neutrophil count ≥1.5×10⁹/L, platelet count ≥60×10⁹/L
   * Liver Function: Total bilirubin ≤1.5× upper limit of normal (ULN), ALT and AST ≤2.5× ULN (≤5× ULN for patients with liver metastasis)
   * Renal Function: Serum creatinine ≤1.5× ULN or creatinine clearance ≥50 mL/min
   * Cardiac Function: Left ventricular ejection fraction ≥40%
9. Informed Consent: The patient or their legal representative has signed the informed consent form.

Exclusion Criteria:

1. Special Types of Sarcoma:

   * Gastrointestinal Stromal Tumor (GIST)
   * Osteosarcoma
   * Ewing's Sarcoma
2. Prior Treatment History:

   * Previous radiotherapy to the same site with a cumulative dose that may exceed the normal tissue tolerance dose
   * Major surgery within 4 weeks
3. Concurrent Diseases:

   * Active autoimmune diseases
   * Diseases requiring systemic immunosuppressive therapy
   * Severe cardiovascular diseases (myocardial infarction, unstable angina, heart failure, etc.)
   * Severe pulmonary diseases (interstitial pneumonia, pulmonary fibrosis, etc.)
   * Active infections requiring systemic anti-infective therapy
4. Central Nervous System Metastasis: Symptomatic brain or spinal metastasis.
5. Pregnancy and Lactation: Women who are pregnant or breastfeeding.
6. Allergy History: Known allergies to the drugs or their components involved in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | week 4

SECONDARY OUTCOMES:
Disease Control Rate | week 4

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No